CLINICAL TRIAL: NCT00006517
Title: Light and Ion Therapy for Seasonal Affective Disorder
Brief Title: Clinical Trials of Three Non-Drug Treatments for Winter Depression (SAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #3032/R01 MH42931-01; R01MH042931-01 (NIH)
Record Dates: First submitted 2000-11-22; First posted 2000-11-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2005-11

CONDITIONS: Seasonal Affective Disorder; Mood Disorders; Depression
Keywords: Seasonal Affective Disorder (SAD); Winter Depression; Mood disorders; Bipolar I and II disorders; Major Depressive Disorder, Recurrent; Light therapy; Phototherapy; Dawn Simulation therapy; Negative air ionization therapy; Chronobiology; Biological rhythms
MeSH Terms: conditions — Seasonal Affective Disorder; Mood Disorders; Depression; Depressive Disorder, Major; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- bright light box (Active Comparator): 30 min exposure shortly after wake-up
  Interventions: Device: bright light box
- high-output negative ion generator (Active Comparator): 90 min exposure prior to wake-up
  Interventions: Device: high-output negative ion generator
- low-output negative ion generator (Placebo Comparator): 90 min exposure prior to wake-up
  Interventions: Device: low-output negative ion generator
- dawn simulator (Active Comparator): naturalistic incremental light exposure 90 min prior to wake-up
  Interventions: Device: dawn simulator
- dawn light pulse (Experimental): rectangular pulse light exposure 13 min before wake-up, matched for total illuminance with dawn signal
  Interventions: Device: dawn light pulse

INTERVENTIONS:
Device: bright light box — 10,000 lux bright light therapy
  Arms: bright light box
Device: dawn simulator — gradual rise in bedroom illumination prior to wake-up
  Arms: dawn simulator
Device: high-output negative ion generator — automated air ion delivery in bedroom prior to wake-up
  Arms: high-output negative ion generator
Device: low-output negative ion generator — automated air ion delivery in bedroom prior to wake-up
  Arms: low-output negative ion generator
Device: dawn light pulse — rectangular light pulse matched for lux.time of dawn simulation delivered prior towake-up
  Arms: dawn light pulse

SUMMARY:
We are offering non-pharmacologic therapy for alleviation of symptoms associated with depressed mood that recurs annually in fall or winter. The treatments are self-administered at home by the patient, with close clinical supervision. Our trials use specially designed devices that replenish two different environmental elements, naturally occurring light and negative ions in the air. Both factors may be reduced in winter, bringing on depression.

DETAILED DESCRIPTION:
The treatments we are investigating include bright light therapy upon awakening, and two contrasting treatments during the final hours of sleep: negative air ionization (provided at two levels) and dawn simulation (also at two levels), both switched on by a silent electronic timer or microprocessor. We hypothesize that the reduced outdoor light availability in winter, as well as reduced concentration of negative ions in the air circulation are both factors that contribute to depression. By supplementing the indoor environment with either ions or light, we are aiming to recreate summer-like conditions that are therapeutic. Our past studies have shown all three methods to have antidepressant effects in patients with seasonal affective disorder (SAD). Unlike light therapy, negative air ionization is imperceptible (you cannot sense when the ionizer is active).

Applications to the program are accepted and reviewed throughout the year. Screening interviews for entry into the program are scheduled between August and February. Patients and researchers both benefit most when applications are received by the start of the individual's "problem season," because this leaves maximum time to explore alternate treatments. Candidates undergo a two-hour personal interview at Columbia-Presbyterian Medical Center that ascertains whether they meet inclusion criteria. At a second two-hour visit we provide a standard medical examination including blood tests, urinalysis and EKG, all without cost. As an alternative, physicals may be performed by one's personal physician. Once the study is underway, there are about five additional one-hour appointments for clinical evaluations, flexibly scheduled during the business day, usually about 10 days apart.

We provide the treatment apparatus on loan. All treatments are scheduled in the morning around the time of awakening. The bedroom treatments (negative ions or dawn simulation) end by the time of awakening. The bright light treatment takes place for half an hour after waking up. Initially, patients are randomly assigned to one of the treatment groups. The treatment must be taken consistently for three weeks at the same time every day, after which it is temporarily suspended to determine whether symptoms return. Given sufficient time within the winter season, patients then have the opportunity to try one of the alternate treatments to determine which works best for them. This provides an informed, confident basis for a treatment plan for subsequent years.

As part of the protocol, patients provide saliva samples on two evenings, which are used to test for the level of melatonin, a hormone that becomes active at night. Results reveal whether a person's internal circadian rhythm is early, late or normal, information that can be used to guide the timing of future treatment. This constitutes a distinct benefit for research participants, since such a diagnostic test is not yet available in medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depression or bipolar disorder, with regular onset of depression in fall or winter and remission in spring
* Able to maintain a regular sleep schedule

Exclusion Criteria:

* Presence of psychiatric disorders other than major depression or bipolar depression
* Current use of antidepressant or recreational drugs, or psychotropic medication or supplements that may affect mood
* Current medical illness or medication that might interfere with response to treatment
* Long-distance travel during the program

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1998-09; Primary Completion 2003-06 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Depression scale score | 3 weeks
  reduction from depressed baseline

SECONDARY OUTCOMES:
time of pineal melatonin onset | 3 weeks
  change from depressed baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Terman, Principal Investigator — Columbia University
Locations (1):
- Columbia Presbyterian Medical Center, New York, New York, United States

REFERENCES:
- [Background] Caldwell M. Mind over time. Discover Magazine, July 1999;50-59. <http://www.discover.com/july_99/featmind.html>
- [Background] Terman M, Lewy AJ, Dijk DJ, Boulos Z, Eastman CI, Campbell SS. Light treatment for sleep disorders: consensus report. IV. Sleep phase and duration disturbances. J Biol Rhythms. 1995 Jun;10(2):135-47. doi: 10.1177/074873049501000206. PMID 7632987
- [Background] Terman M, Terman JS, Ross DC. A controlled trial of timed bright light and negative air ionization for treatment of winter depression. Arch Gen Psychiatry. 1998 Oct;55(10):875-82. doi: 10.1001/archpsyc.55.10.875. PMID 9783557
- [Background] Terman M; Terman JS; Williams JBW. Seasonal affective disorder and its treatments. J Pract Psychiatry Behav Health 1998;5:387-303. <http://www.practicalpsychiatry.com>
- See also: Click here for more information about our study. Also, you can print out a confidential preliminary application to mail or fax to our center for quick review. — http://www.columbiapsychiatry.org/cs/cltbr.html
- See also: Click here for information about SAD and its treatments, presented by the Center for Environmental Therapeutics, a 501(c)(3) nonprofit professional agency. — http://www.cet.org/
- See also: Background reference: Click hear to read the abstract of Dr. Terman's article, "Seasonal Affective Disorder and its Treatments," in the Journal of Practical Psychiatry and Behavioral Health (at the site, click on "Contents," September 1998). — http://www.practicalpsychiatry.com/